CLINICAL TRIAL: NCT04946565
Title: The Impact of Sinopharm COVID-19 Vaccination on Male Fertility of the Egyptian Population
Brief Title: The Impact of Sinopharm COVID-19 Vaccination on Male Fertility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Tarek Anis, Professor of Andrology, Cairo University
Other Study IDs: TBA
Record Dates: First submitted 2021-06-28; First posted 2021-07-01 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Male Infertility; Hypogonadism, Male
MeSH Terms: conditions — Infertility, Male; Eunuchism | interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sinopharm vaccine group: Participants scheduled to receive the Sinopharm vaccine will be evaluated on its effect on semen parameters for up to 6 months post vaccination.
  Interventions: Diagnostic Test: Semen analysis

INTERVENTIONS:
Diagnostic Test: Semen analysis — Semen analysis according to WHO laboratory manual for the examination and processing of human semen, Fifth edition

SUMMARY:
The investigators shall study the effect of Sinopharm vaccination on semen parameters and serum testosterone

DETAILED DESCRIPTION:
The investigators shall compare semen parameter (sperm density, sperm motility, and percentage of abnormal sperm form) as well as morning serum testosterone before vaccination, and 3 months after the second dose of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

Receiving Sinopharm COVID-19 vaccines Male age 18-50 years old

Exclusion Criteria:

* Adults unable to consent
* Men who have been receiving Testosterone replacement therapy or anabolic steroids within the last year
* Men with a history of male infertility
* Men with a genetic or other medical condition known to be associated with decreased semen parameters Positive COVID-19 PCR test within the 3 months

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men of reproductive age scheduled for COVID-19 Sinopharm Vaccine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Sperm density count/ml | up to 6 months
  As measured from semen samples
Total sperm count per ejaculate | up to 6 months
  As measured from semen samples
Percentage of motile sperm | up to 6 months
  As measured from semen samples
Percentage of abnormal sperm forms | up to 6 months
  As measured from semen samples

SECONDARY OUTCOMES:
Morning serum testosterone | up to 6 months
  Total serum testosterone measured using immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tarek H Anis, M.D., Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt